CLINICAL TRIAL: NCT03315286
Title: Validation of SHADE a Mobile Technology for Monitoring of Ultraviolet Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: YouV Labs Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1609017593; HHSn261201700005c (Other: National Institute of Health)
Record Dates: First submitted 2017-10-11; First posted 2017-10-20 (Actual); Results first posted 2019-11-07 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Skin Cancer; Actinic Keratoses; Ultraviolet-Induced Change in Normal Skin; Behavior, Health; Behavior, Risk Reduction
Keywords: ultraviolet light; dosimetry; actinic keratosis; skin cancer; sun counseling; wearable device
MeSH Terms: conditions — Skin Neoplasms; Keratosis, Actinic; Health Behavior; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Device: SHADE Ultraviolet Sensor (Experimental): Patients will receive an Ultraviolet (UV) sensor that will quantify their UV exposure through a linked smartphone application. Patients will also receive clinical counseling by their dermatologist regarding sun protection and avoidance
  Interventions: Device: SHADE Ultraviolet Sensor; Behavioral: Standard of care counseling
- Standard of Care Counseling (Active Comparator): Patients will receive clinical counseling by their dermatologist regarding sun protection and avoidance
  Interventions: Behavioral: Standard of care counseling

INTERVENTIONS:
Device: SHADE Ultraviolet Sensor — Patients will wear device for 6 months in addition to their own method of photo-protection.
  Other Names: SHADE
  Arms: Device: SHADE Ultraviolet Sensor
Behavioral: Standard of care counseling — Patients will use their own method of photo-protection

SUMMARY:
This study will evaluate the safety and effectiveness of Shade for the management of UV-induced skin complications and data collected from this study will be used to support the proposed indications for use.

DETAILED DESCRIPTION:
The incidence of non-melanoma skin cancers, due to increased ultraviolet (UV) exposure, has increased by 300% over the past 2 decades. The innovative UV sensor, Shade, is designed to help people manage their UV exposure by quantifying their UV exposure levels through a linked smartphone application. In order to validate the effectiveness of Shade, we propose conducting a study communicating the level of UV exposure and correlating it with the development of actinic keratosis (AK), a precancerous lesion of the skin. We will recruit patients with multiple repeat AK's, as this population continues to develop AKs every year. We will include renal transplant patients. The risk of developing squamous cell carcinoma (SCC) in renal transplant patients is 65 times higher than normal patients. They are an ideal patient population for this study. We will evaluate the UV monitor's effectiveness in decreasing the number of AKs over a summer. This randomized partially blinded study will recruit 120 patients with a recent history of AK lesions and evaluate the incidence of new AKs after one summer. We will perform a control versus study group analysis. Half of the subjects (study group) will be randomly assigned to use the sensor along with its smartphone application, while the other half (control group) will receive standard of care treatment involving counseling to avoid sun exposure. Subjects will have regular standard of care visits with the dermatologist who will follow the number of actinic keratosis via clinical exam and photography. The primary outcome will be a statistically significant reduction by at least 25% of the cumulative number of newly occurred AK lesions between the control and the study group over one summer, counted at enrollment and follow-up. In subjects at one study site, skin DNA damage will also be assessed using cyclobutane pyrimidine dimers (CPD) levels measured by ELISA in both sun exposed (cheek) and sun protected skin (buccal mucosa) in both the study and control groups. Secondary outcomes will look at clinical decreases by 25% in CPD levels after using the sensor.

ELIGIBILITY:
Inclusion Criteria:

* between 18-80 years of age
* given a diagnosis of actinic keratosis in the past year and/or has had a history of >5 actinic keratosis over the past 5 years
* has a compatible smartphone ((Apple version >= 7, Android version >= 4.4.2; no Jitterbug or Samsung Galaxy J3)
* willing to commit to dermatology visits (including standard of care visits) every 3 months for 6 months

Exclusion Criteria:

* received UV therapy within the past 6 months
* work/lifestyle incompatible with wearing a UV sensor over the course of 1 year
* has difficulty controlling UV exposure
* has a medical condition judged incompatible with the study by the enrolling physician including the presence of an ICD or an existing plan for extended inpatient treatment
* has received field therapy (i.e., entire face or scalp) for the treatment of actinic keratosis (i.e., topical imiquimod, 5-fluorouracil, photodynamic therapy) in the past 3 months
* is an employee or direct relative of an employee of the investigational site or study sponsor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Varghese, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be available through publications, presentations at scientific symposia and seminars. Efforts will be made to publish our research findings in scientific journals. All final peer-reviewed manuscripts that arise from this proposal will be submitted to the digital archive PubMed Central. To encourage use of the data, subject level device data will be made available on request to qualified researchers including to NIH staff who agree to restrictions against public release of the data, attempts to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on the redistribution of the data to third parties, and proper acknowledgement of the data resource.
Supporting Information: Study Protocol
Time Frame: 1-5 years
Access Criteria: Requests will be made directly to SHADE by email through contact information to be provided on its web site and included in each publication based on these data. These data will be shared without fee through a single use web link which will enable the secure download of subject level device data in .csv format.

REFERENCES:
- [Derived] Dumont ELP, Kaplan PD, Do C, Banerjee S, Barrer M, Ezzedine K, Zippin JH, Varghese GI. A randomized trial of a wearable UV dosimeter for skin cancer prevention. Front Med (Lausanne). 2024 Mar 1;11:1259050. doi: 10.3389/fmed.2024.1259050. eCollection 2024. PMID 38495115

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 14 patients with kidney transplantation & actinic keratosis from 10/2018 to 4/2018. We recruited another 97 patients with only a history of actinic keratosis without a history of kidney transplantation between 4/2018 and 7/2018. Patient were all recruited at one academic institution. We are presenting the data of the 97 patients.
Period: Overall Study
Arm/Group | Device: SHADE Ultraviolet Sensor | Standard of Care Counseling
Started | 50 | 47
Completed | 49 | 43
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: We are posting the results of patients without a transplant (97).
Groups:
- Total: Total of all reporting groups
Arm/Group | Device: SHADE Ultraviolet Sensor | Standard of Care Counseling | Total
Number analyzed (Participants) | 50 | 47 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 12 | 37
  >=65 years | 25 | 35 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 20 | 34
  Male | 36 | 27 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 45 | 47 | 92
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 49 | 47 | 96
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 50 | 47 | 97
Baseline measurement of Actinic keratosis [Mean (Full Range); unit: lesions] — Population: We measured only the non transplant patients (97). 14 were excluded from baseline analysis.
  lesions | 6.42 [0 to 36] | 6.212 [0 to 25] | 6.319 [0 to 36]

OUTCOME MEASURES:

1. Primary Outcome: Quantification of Actinic Keratosis Using the UV Sensor vs. Control Group
Description: Clinical counting of new actinic keratosis at 3 month intervals for a total duration of 6 months. Patient's actinic keratosis were counted at baseline (0 months), 3 months and 6 months. The average number of actinic keratosis at 6 months is only reported.
Time Frame: 6 months
Population: We are posting the results of patients without a transplant (97). Out of the 97 subjects, in the device group, 49 subjects completed the study. 1 subject was removed for protocol violation. In the control group, 43 subjects completed the study, 3 subjects were lost to follow up and 1 subject was removed for protocol violation.
Measure: Mean (Full Range); unit: lesions
Arm/Group | Device: SHADE Ultraviolet Sensor | Standard of Care Counseling
Number analyzed (Participants) | 49 | 43
lesions | 4.53 [0 to 14] | 4.74 [0 to 22]
Statistical Analysis 1: Comparison: Device: SHADE Ultraviolet Sensor vs Standard of Care Counseling; Test type: Superiority; p = 0.8, t-test, 2 sided

2. Secondary Outcome: Quantification of Non Melanoma Skin Cancers After Using the UV Sensor vs. Control Group
Description: Clinical counting of new non melanoma skin cancers at 3 month intervals for a total duration of 6 months. Patient's non melanoma skin cancers were counted at baseline (0 months), 3 months and 6 months. The average number of non melanoma skin cancers at 6 months is only reported.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Full Range); unit: lesions
Arm/Group | Device: SHADE Ultraviolet Sensor | Standard of Care Counseling
Number analyzed (Participants) | 49 | 43
lesions | 0.04 [0 to 1] | 0.232 [0 to 2]
Statistical Analysis 1: Comparison: Device: SHADE Ultraviolet Sensor vs Standard of Care Counseling; Test type: Superiority; p = 0.03, t-test, 2 sided

3. Secondary Outcome: Impact of UV Sensor (SHADE) on Patient's Quality of Life as Measured by PROMIS - Depression
Description: PROMIS (Patient-Reported Outcomes Measurement Information System) surveys will be given to patients at at baseline (0 months), 3 months and 6 month . Specifically we will include questions about anxiety, depression, and ability to participate in social roles and activities. The surveys will be scored on a scale of 1 to 5. 1 indicates never, 5 indicates always. An example of a question would be "I felt fearful" and the patient would score this question on a scale of 1-5 as indicated above. The results are scored using item-level calibrations via HealthMeasures.net Scoring Service. The total raw score (aggregate of the scores) is rescaled into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10.
Time Frame: Baseline, 3 months and 6 months. data at baseline and 6 months will be reported
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Device: SHADE Ultraviolet Sensor | Standard of Care Counseling
Number analyzed (Participants) | 49 | 43
units on a scale
  baseline | 44.2 [38 to 62] | 43.6 [38 to 55]
  6 months | 45.3 [38 to 62] | 43.7 [38 to 59]
Statistical Analysis 1: Comparison: Device: SHADE Ultraviolet Sensor vs Standard of Care Counseling; Baseline results are reported here; Test type: Superiority; p = 0.6, t-test, 2 sided
Statistical Analysis 2: Comparison: Device: SHADE Ultraviolet Sensor vs Standard of Care Counseling; 6 month data is reported here; Test type: Superiority; p = 0.3, t-test, 2 sided

4. Secondary Outcome: Impact of UV Sensor (SHADE) on Patient's Quality of Life as Measured by PROMIS - Anxiety
Description: as for outcome 3
Time Frame: Baseline, 3 months and 6 months. data at baseline and 6 months will be reported
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Device: SHADE Ultraviolet Sensor | Standard of Care Counseling
Number analyzed (Participants) | 49 | 43
units on a scale
  baseline | 46.2 [37 to 63] | 44.1 [37 to 65]
  6 months | 46.3 [37 to 66] | 44.7 [37 to 63]
Statistical Analysis 1: Comparison: Device: SHADE Ultraviolet Sensor vs Standard of Care Counseling; Baseline data is reported here; Test type: Superiority; p = 0.2, t-test, 2 sided
Statistical Analysis 2: Comparison: Device: SHADE Ultraviolet Sensor vs Standard of Care Counseling; 6 month data is reported here; Test type: Superiority; p = 0.4, t-test, 2 sided

5. Secondary Outcome: Impact of UV Sensor (SHADE) on Patient's Quality of Life as Measured by PROMIS - Ability to Participate in Social Roles and Activities
Description: as for outcome 3
Time Frame: Baseline, 3 months and 6 months. data at baseline and 6 months will be reported
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Device: SHADE Ultraviolet Sensor | Standard of Care Counseling
Number analyzed (Participants) | 49 | 43
units on a scale
  baseline | 57 [34 to 65] | 60 [44 to 65]
  6 months | 55.8 [36 to 65] | 62.1 [47 to 65]
Statistical Analysis 1: Comparison: Device: SHADE Ultraviolet Sensor vs Standard of Care Counseling; baseline data is reported here; Test type: Superiority; p = 0.07, t-test, 2 sided
Statistical Analysis 2: Comparison: Device: SHADE Ultraviolet Sensor vs Standard of Care Counseling; 6 month data is reported here; Test type: Superiority; p = 0.0002, t-test, 2 sided

6. Secondary Outcome: Quantification of Melanoma Skin Cancers After Using the UV Sensor vs. Control Group
Description: Clinical counting of new non melanoma skin cancers at 3 month intervals for a total duration of 6 months. Patient's melanoma skin cancers were counted at baseline (0 months), 3 months and 6 months. The number of melanoma skin cancers at each time point is reported.
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: lesions
Arm/Group | Device: SHADE Ultraviolet Sensor | Standard of Care Counseling
Number analyzed (Participants) | 49 | 43
lesions
  baseline | 0 | 1
  3 months | 0 | 1
  6 months | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse effects were evaluated over the course of the study which was 6 months.
Description: All adverse reports were reported using an adverse event case report form. These are reported immediately into the patient's file and reported to the IRB.
Arm/Group | Device: SHADE Ultraviolet Sensor | Standard of Care Counseling
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/47
Other Adverse Events (participants affected / at risk) | 0/50 | 0/47

LIMITATIONS AND CAVEATS:
Transplant patient population was limited, too small a size. Ideally, we would have liked to monitor patients over 1 year.

Secondary outcomes of melanomas:, could not power the statistical analysis due to small number of diagnosed melanomas.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT03315286/Prot_SAP_000.pdf